CLINICAL TRIAL: NCT07348055
Title: A Phase Ib/IIa Clinical Trial Evaluating the Safety, Tolerability, and Efficacy of GR1803 Injection in Subjects With Systemic Lupus Erythematosus
Brief Title: A Study of GR1803 in Systemic Lupus Erythematosus
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genrix (Shanghai) Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GR1803-007
Record Dates: First submitted 2025-12-25; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Systemic Lupus Erthematosus; Auto Immune Disease
Keywords: BCMA/CD3 Bispecific Antibody; systemic lupus erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GR1803 injection dose 1 (Experimental)
  Interventions: Biological: GR1803 injection
- GR1803 injection dose 2 (Experimental)
  Interventions: Biological: GR1803 injection
- GR1803 injection dose 3 (Experimental)
  Interventions: Biological: GR1803 injection
- GR1803 injection dose 4 (Experimental)
  Interventions: Biological: GR1803 injection

INTERVENTIONS:
Biological: GR1803 injection — step-up dosing, Dose and frequency according to the protocol

SUMMARY:
to evaluate the safety and efficacy of GR1803 in the treatment of patients with systemic lupus erythematosus

ELIGIBILITY:
Inclusion Criteria:

* comfirmed diagnosis of systemic lupus erythematosus
* SLEDAI-2K≥6分
* written informed consent and ability to comply with protocol requirements
* have received adequate dose of glucocorticoids, antimalarials, immunosuppressants for 3 months

Exclusion Criteria:

* with unstable acute and chronic diseases
* active infection
* history of malignant tumor within 5 years

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
incidence of adverse event | 52 week
  incidence of adverse event

SECONDARY OUTCOMES:
efficacy of GR1803 | 52 week
  clinical response of SLE

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided